CLINICAL TRIAL: NCT04282993
Title: Wearable Devices for Secondary Prevention of Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Di Lazzaro Vincenzo, Head of Neurology, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AN01
Record Dates: First submitted 2020-02-19; First posted 2020-02-25 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Stroke, Ischemic; Atrial Fibrillation
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation | interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wearable Devices Monitoring (Experimental): Patients will be provided with wearable devices for at-home monitoring heart rhythm and rate, blood pressure, pulse oximetry, quality and quantity of sleep, and pace counting.
  Interventions: Device: Wearable devices for identifying and measuring risk factors for ischemic stroke
- Standard of Care Monitoring (Active Comparator): Patients will be evaluated by periodical clinical visits.
  Interventions: Other: Standard of care monitoring

INTERVENTIONS:
Device: Wearable devices for identifying and measuring risk factors for ischemic stroke — Identifying and monitoring cerebrovascular risk factors using wearable devices
  Arms: Wearable Devices Monitoring
Other: Standard of care monitoring — Periodical medical examinations
  Arms: Standard of Care Monitoring

SUMMARY:
Ischemic stroke is an important cause of death and disability in Western countries. Different risk factors have been identified such as hypertension, diabetes, dyslipidemia, smoke, atrial fibrillation, obesity, and sedentary. The aim of this study is to evaluate the feasibility of an approach based on the use of wearable devices for the identification and reduction of risk factors in patients with previous history of ischemic stroke or transient ischemic attack.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal 50 years
* Recent transient ischemic attack or minor stroke

Exclusion Criteria:

* Patients with significant cognitive impairment
* Patients dependent in the instrumental activities of daily life
* Patients not able to respect the frequency of monitoring program
* Patients with history of atrial fibrillation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Compliance of patients to at-home follow-up by means of wearable devices | 1 month
  Number of measurements actually performed in comparison to number of expected measurements

SECONDARY OUTCOMES:
Atrial fibrillation Detection Rate | 1 month
  Percentage of subjects with atrial fibrillation detected within 1 month of follow-up
Prevalence of Recurrent Stroke or Transient Ischemic Attack | 1 month
  Prevalence of subjects with recurrent stroke or Transient Ischemic Attack within 1 month of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Di Lazzaro, MD, Principal Investigator — Campus Bio-Medico University
Locations (1):
- Università Campus Bio-Medico di Roma, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No